CLINICAL TRIAL: NCT02259413
Title: Effect of an Exercise Rehabilitation Program on Symptom Burden and Quality of Life in Hemodialysis: A Randomized Controlled Study
Brief Title: Effect of an Exercise Rehabilitation Program on Symptoms in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The Wellness Institute at Seven Oaks General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2014:088
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: End-stage Renal Disease; Renal Failure Chronic Requiring Hemodialysis
Keywords: Hemodialysis; End-stage renal disease; Exercise; Symptom Burden
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Rehabilitation (Experimental): Participants will receive baseline exercise counselling as per Standard Care group. Participants will then participate in a 26-week exercise rehabilitation program incorporating 3 components:
  1. One-to-one self-management/resistance education once per week during the first 4 weeks of intervention. Participants will subsequently receive resistance training material to allow for home exercise for the remaining 22 weeks of the intervention.
  2. Intradialytic aerobic exercise on a cycle ergometer 3 times weekly for 26 weeks at their usual hemodialysis sessions.
  3. Four additional one-to-one standardized education sessions will be completed during the intervention period.
  Interventions: Behavioral: Exercise Rehabilitation
- Standard Care (No Intervention): Participants will receive one exercise counseling session as part of their baseline assessment. Participants in the control group will not undergo any other exercise counseling or formal exercise intervention, but will not be prohibited from participating in exercise outside of the study protocol.

INTERVENTIONS:
Behavioral: Exercise Rehabilitation — This intervention will consist of lifestyle education, home-based resistance exercise and stationary cycling during hemodialysis sessions. Duration of the intervention will be 26 weeks
  Arms: Exercise Rehabilitation

SUMMARY:
The purpose of this study is to determine whether participation in a 26-week exercise rehabilitation program is effective at reducing symptom burden and improving quality of life in individuals receiving chronic hemodialysis.

DETAILED DESCRIPTION:
Individuals with end-stage kidney disease requiring HD suffer from multiple symptoms, which have limited effective treatments. Symptom burden, the combined impact of number and severity of symptoms, negatively impacts functional status and health-related quality of life (HRQOL) in HD. Small interventional trials suggest exercise can mitigate specific individual symptoms, but impact of exercise on overall symptom burden in HD is unknown. Dialysis patients have identified improving symptom burden and HRQOL as research priorities. We propose the first randomized controlled trial (RCT) investigating the effect of exercise rehabilitation on symptom burden in individuals on HD.

Hypothesis: In individuals on HD, participation in a 26-week exercise rehabilitation (rehab) program will reduce symptom burden and improve HRQOL, resulting in reduced disability and improved long-term clinical outcomes as compared with standard care.

Study Design: Single-centre RCT with one-to-one parallel design, allocation concealment and assessor blinding

Study Population: Adults receiving chronic in-centre HD for > 3 months with at least one dialysis-related symptom; n=150

Intervention: Standard care plus 26-week structured rehab program (lifestyle education, resistance exercise and cycling during HD).

Control: Standard care (baseline exercise counseling)

Outcomes measured at baseline, 12, 26 and 52 weeks.

Data Analysis: Will be performed on an intention to treat, available case basis with t-tests or Mann Whitney U for continuous outcomes, as per data distribution and Chi square tests for categorical outcomes. Mixed effects modeling will account for repeated outcome measures over time. Poisson regression will be performed for hospitalization analysis.

Anticipated Outcomes: Mean symptom burden severity score will decrease by 20% from baseline in the intervention group at 12 weeks. Due to sustained physical activity in the intervention group, symptom burden will remain lower in this group at 6 months. In contrast, the control group will see no improvement in symptom burden from baseline.

ELIGIBILITY:
Inclusion Criteria:

* greater than 3 months after starting chronic hemodialysis
* no planned change in hemodialysis modality or relocation outside of Winnipeg during study intervention period (26 weeks)
* assessed to be safe and able to exercise by HD unit nephrologist
* ability to communicate in English and provide informed written consent

Exclusion Criteria:

* acute coronary syndrome in past 3 months
* unstable arrhythmia
* shortness of breath at rest or with minimal activity (NYHA Class 4)
* symptomatic hypoglycaemia (> 2x/week in week prior to enrolment)
* currently participating in the Manitoba Renal Program clinical intradialytic cycling program
* score of 0 on Dialysis Symptom Index when administered at time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Change in dialysis symptom burden at 12 weeks | Measured at study baseline and 12 weeks after study start
  Measured using change in the Dialysis Symptom Index

SECONDARY OUTCOMES:
Change in dialysis symptom burden at 26 and 52 weeks | Measured at study baseline, 26 and 52 weeks after study start
  Measured using change in the Dialysis Symptom Index
Change in modified symptom burden | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured using change in modified Dialysis Symptom Index
Change in health-related quality of life | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured by self-report using the EuroQol 5D-5L (EQ5D-5L) and EuroQol Visual Analogue Scale.
Change in time for recovery post-dialysis | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured in minutes with the question "Approximately how much time does it take to recover from a dialysis session"
Change in endurance/exercise capacity | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured using the Incremental Shuttle Walk Test
Change in frailty status | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured using the Modified Fried Criteria for frailty.
Change in self-efficacy for exercise | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured using the Self-Efficacy for Exercise Survey a 9 item self-reported assessment tool

OTHER OUTCOMES:
Change in physical activity behaviour pattern | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured in 2 ways:
  1. Subjectively using the self-reported Godin-Shephard Leisure Time Physical Activity Questionnaire
  2. Objectively using multi-directional accelerometers (Actical Physical Activity Monitors TM) which will be worn for 7 days at each measurement time point
  2.
Hospitalization rate | Measured at study baseline, 12, 26 and 52 weeks after study start
  Measured by number of hospitalizations and length of stay for each hospitalization
Mortality | Measured at 1 year after starting dialysis
  Measured as the proportion of people who died during the first year on dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Clara J Bohm, MD, MPH, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - Health Sciences Centre, Winnipeg, Manitoba
  - Seven Oaks General Hospital, Winnipeg, Manitoba
  - St. Boniface Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Protocol Publication — http://pmc.ncbi.nlm.nih.gov/articles/PMC10993676/pdf/10.1177_20543581241234724.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Formal protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT02259413/Prot_SAP_003.pdf
  • Informed Consent Form (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT02259413/ICF_001.pdf